CLINICAL TRIAL: NCT01408290
Title: A Randomized, Double Blind, Multicentre Study to Evaluate Safety and Immunogenicity of Four Fluval AB-Like Influenza Vaccines With 3.5 μgHA, 6 μgHA, 9 μgHA Or 15 μgHA Of A/H1N1, A/H3N2 and B Influenza Antigens in Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity Study of Fluval AB-Like Flu Vaccines With 3.5, 6, 9 or 15 μg HA in Adult and Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FluvalAB-H-14; 2011-003166-32 (EudraCT Number)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Influenza
Keywords: seasonal; prevention; influenza; infection; influenza vaccine; vaccine; influenza in humans
MeSH Terms: conditions — Influenza, Human; Infections | interventions — Vaccination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- FAB-6011 (Experimental): - One 0.5 mL injection of FAB-6011 trivalent influenza vaccine containing 6μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens (32 subjects aged 18-60 years /Group 2A/ and 32 subjects aged over 60 years /Group 2E/).
  Interventions: Biological: Vaccination with FAB-6011
- FAB-9011 (Experimental): - One 0.5 mL injection of FAB-9011 trivalent influenza vaccine containing 9μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens (32 subjects aged 18-60 years /Group 3A/ and 32 subjects aged over 60 years/Group 3E/).
  Interventions: Biological: Vaccination with FAB-9011
- FLUVALAB (Experimental): - One 0.5 mL injection of FLUVAL AB trivalent influenza vaccine containing 15μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens (32 subjects aged 18-60 years /Group 4A/ and 32 subjects aged over 60 years/Group 4E/).
  Interventions: Biological: Vaccination with FluvalAB
- FAB-3511 (Experimental): - One 0.5 mL injection of FAB-3511 trivalent influenza vaccine containing 3.5μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens (32 subjects aged 18-60 years /Group 1A/ and 32 subjects aged over 60 years /Group 1E/).
  Interventions: Biological: Vaccination with FAB-3511

INTERVENTIONS:
Biological: Vaccination with FAB-3511 — One 0.5 mL injection of FAB-3511 trivalent influenza vaccine containing 3.5μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens.
  Other Names: FAB-3511
  Arms: FAB-3511
Biological: Vaccination with FAB-6011 — One 0.5 mL injection of FAB-6011 trivalent influenza vaccine containing 6μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens.
  Other Names: FAB-6011
  Arms: FAB-6011
Biological: Vaccination with FAB-9011 — One 0.5 mL injection of FAB-9011 trivalent influenza vaccine containing 9μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens.
  Other Names: FAB-9011
  Arms: FAB-9011
Biological: Vaccination with FluvalAB — One 0.5 mL injection of FLUVAL AB trivalent influenza vaccine containing 15μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens.
  Other Names: FluvalAB
  Arms: FLUVALAB

SUMMARY:
The purpose of this study is to determine the immunogenicity, tolerability and dose-effect relationship of one 0.5 mL intramuscular (IM) injection of four FLUVAL AB-like trivalent influenza vaccines containing either 3.5μgHA, 6μgHA,9μgHA or 15μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens in adults and elderly people.

DETAILED DESCRIPTION:
Primary immunogenicity objectives

* To assess immunogenicity of one 0.5 mL intramuscular (IM) injection of four FLUVAL AB-like trivalent influenza vaccines containing either 3.5μgHA, 6μgHA, 9μgHA or 15μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens, as measured by haemagglutination inhibition (HI) test 21 days after vaccination in compliance with the requirements of the current European Union recommendations as determined in CPMP/BWP/214/96.
* To determine dose-effect relationship between one 0.5 mL IM injection of four FLUVAL AB-like trivalent influenza vaccines containing either 3.5μgHA, 6μgHA, 9μgHA or 15μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens and immune response provoked 21 days after vaccination in terms of pre- and postimmunization HA titers as measured by HI test.

Secondary immunogenicity objectives

* To assess immunogenicity of one 0.5 mL IM injection of four FLUVAL AB-like trivalent influenza vaccines containing either 3.5μgHA, 6μgHA, 9μgHA or 15μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens, as measured by HI test 14 days after vaccination in compliance with the requirements of the current European Union recommendations as determined in CPMP/BWP/214/96.
* To find the highest dose of FLUVAL AB-like trivalent influenza vaccine among 3.5μgHA, 6μgHA and 9μgHA the response of which differs from that of dose 15μgHA in terms of post-immunization HA titers as measured by HI test 21 days after vaccination.
* To find the highest dose of FLUVAL AB-like trivalent influenza vaccine among 3.5μgHA, 6μgHA and 9μgHA the response of which differs from that of dose 15μgHA in terms of post-immunization HA titers as measured by HI test 14 days after vaccination.
* To find the highest dose of FLUVAL AB-like trivalent influenza vaccine among 3.5μgHA, 6μgHA and 9μgHA the response of which differs from that of dose 15μgHA in terms of the percentage of subjects achieving seroconversion or significant increase in antibody titer at day 21 after vaccination.
* To find the highest dose of FLUVAL AB-like trivalent influenza vaccine among 3.5μgHA, 6μgHA and 9μgHA the response of which differs from that of dose 15μgHA in terms of the percentage of subjects achieving seroconversion or significant increase in antibody titer at day 14 after vaccination.
* To find the highest dose of FLUVAL AB-like trivalent influenza vaccine among 3.5μgHA, 6μgHA and 9μgHA the response of which differs from that of dose 15μgHA in terms of Day 21/Day 0 geometric mean titer ratios (GMTRs) as determined by HI.
* To find the highest dose of FLUVAL AB-like trivalent influenza vaccine among 3.5μgHA, 6μgHA and 9μgHA the response of which differs from that of dose 15μgHA in terms of Day 14/Day 0 geometric mean titer ratios (GMTRs) as determined by HI.

Safety and tolerability objective

* To evaluate the safety of the administration of one 0.5 mL IM injection of four FLUVAL AB-like trivalent influenza vaccines containing either 3.5μgHA, 6μgHA,9μgHA or 15μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens.

ELIGIBILITY:
Inclusion Criteria:

* male and female adult volunteers aged 18 years or older,
* mentally competent,
* able to understand and comply with all study requirements,
* willing and able to give written informed consent prior to initiation of study procedures,
* in good health (as determined by clinical judgement of the investigator on the basis of medical history and existing medical condition) or are in stable medical condition. Subjects will not be excluded with known, adequately treated, clinically significant organ or systemic diseases (e.g. asthma or diabetes), such that, in the opinion of the investigator, the significance of the disease will not compromise the subject's participation in the study.
* Female subjects aged 18 to 60 years (i.e. participants of childbearing potential) with a negative result from the urine pregnancy test prior to vaccination who agrees to use an acceptable contraception method or abstinence throughout the trial and not become pregnant for the duration of the study.
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Pregnancy, breast-feeding or positive urine pregnancy test at baseline prior to vaccination. Female subjects who are able to bear children but not willing to use an acceptable contraception method for the duration of the study.
* Hypersensitivity to eggs, chicken protein, thiomersal, formaldehyde, gentamycin, ciprofloxacin, neomycin or any other component of the vaccine;
* History of anaphylactic shock or neurological symptoms or signs following administration of any vaccine;
* History of Guillain-Barré syndrome;
* Serious disease, such as cancer, autoimmune disease, advanced arteriosclerotic disease, complicated diabetes mellitus, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure;
* Immunosuppressive therapy within the past 36 months;
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids;
* Receipt of immunostimulants;
* Receipt of parenteral immunoglobulin, blood products and/or plasma derivates within the past 3 months;
* Suspected or known HIV, HBV or HCV infection;
* Acute disease and/or axillary temperature ≥37oC within the past 3 days;
* Vaccine therapy within the past 4 weeks;
* Influenza vaccination (any kind) within the past 6 months;
* Experimental drug therapy within the past 4 weeks;
* Concomitant participation in another clinical study;
* Any condition which, in the opinion of the investigator, may interfere with the evaluation of the study;
* Past or current psychiatric disease of the subject that upon judgement of the investigator may have effect on the objective decision-making of the subject;
* Alcohol or drug abuse of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
MEASURES OF IMMUNOGENICITY | 21-28 days following vaccination
  The measures of immunogenicity, for all evaluable subjects by using HI test are:
  * the GMTs at Day 0, at Day 14 and at Day 21 as determined by HI;
  * the Day 14/Day 0, the Day 21/Day 0 and the Day 21/Day 14 geometric mean titer ratios (GMTRs) as determined by HI;
  * the percentage of subjects achieving seroconversion1 or significant increase in antibody titer2 at Day 14 an at Day 21, as determined by HI;
  * the percentage of subjects achieving a titer ≥40 at Day 0, at Day 14 and at Day 21 as determined by HI.

SECONDARY OUTCOMES:
MEASURES OF SAFETY | 21-28 days following vaccination
  * Number and percentage of subjects with at least one local reaction between Day 0 and Day 7 after vaccination.
  * Number and percentage of subjects with at least one systemic reaction between Day 0 and Day 7 after vaccination.
  * Number and percentage of subjects with at least one adverse event between Day 0 and the study termination visit at Day 21.

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Kollar, MD, Study Director — Omninvest Ltd; József Fűzi, MD, Principal Investigator — Family Doctor's Office, Dunakeszi; Ágnes Hasitz, MD, Principal Investigator — Family Doctor's Office, Szentendre; Judit Simon, MD, Principal Investigator — Family Doctor's Office, Budapest; Péter Torzsa, MD, Principal Investigator — Family Doctor's Office, Budapest
Locations (3):
- Hungary (3):
  - Family Doctor's Office, Dunakeszi, Pest County
  - Family Doctor's Office, Szentendre, Pest County
  - Family Doctor's Office, Budapest